CLINICAL TRIAL: NCT04445077
Title: Effects of a Competency-based Education Program on Care Home Staff's Sense of Competence Related to Dementia Care in Mainland China: A Mixed-methods Approach
Brief Title: Education Program for Care Home Staff
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yayi ZHAO, Principal Investigator, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019.500
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Dementia
Keywords: dementia; long-term care; competency; education; staff
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The education will be delivered weekly with 60-90 minutes per lecture for eight lectures. Multiple teaching methods will be used, including lectures, structured handouts, video, role play, case study and discussion. During the study period, the research team will provide ongoing support and consultation through electronic communication and bimonthly field visits.
  Interventions: Other: Dementia Competence Education for care home setting
- Control group (Other): Printed materials will be given to the participants in the control group for their self-study.
  Interventions: Other: Printed educational materials

INTERVENTIONS:
Other: Dementia Competence Education for care home setting — The intervention is a competency-based education program for care home staff who provide dementia care in Mainland China.
  Arms: Intervention group
Other: Printed educational materials — The educational materials will be delivered to the participants in the control group for their self-study.
  Arms: Control group

SUMMARY:
The competence of care home staff in dementia care is highly influential to the quality of care that adversely affects both people living with dementia and staff and in Mainland China where knowledge on dementia among care home staff was generally poor and this area is under-researched. This study aims at developing a competency-based culturally-sensitive education program on dementia care for care home staff through literature review, qualitative study. And then a quasi-experiment design without random assignment will be conducted to evaluate the effects of this program on care home staff's sense of competence, knowledge, attitudes, and care approach related to dementia care and staff satisfaction with the intervention. Focus group interviews will be conducted to understand participants' experience about the education program after the intervention. This study is expected to provide an effective way to improve care homes staff's competence in dementia care thereby improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

Care homes:

* having at least 10 people with dementia living in;
* with at least 10 care staff working for people with dementia;
* which do not have any educational activities for staff in dementia three months before the study and staff training plan during the whole study period;
* whose management level agrees to participate.

Care staff:

* working for people with dementia;
* speaking and reading Chinese;
* being willing to participate in the study.

Exclusion Criteria:

* having any educational activities in dementia three months before the study;
* having a training plan during the whole study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change of sense of competence in dementia care | Sense of competence in dementia care changes from baseline to immediately after intervention (2 months).
  Sense of competence in dementia care will be measured by Sense of Competence in dementia care scale.The total score is 17-68 by adding up the score of each item. Higher scores mean higher level of sense of confidence.
Change of Sense of competence in dementia care | Sense of competence in dementia care changes from immediately after intervention to three months after intervention.
  Sense of competence in dementia care will be measured by Sense of Competence in dementia care scale.The total score is 17-68 by adding up the score of each item. Higher scores mean higher level of sense of confidence.

SECONDARY OUTCOMES:
Change of knowledge on dementia | Knowledge on dementia changes from baseline to immediately after intervention (2 months).
  Knowledge on dementia will be assessed by using Dementia Knowledge Assessment Scale. The total score is 0 to 50 by adding up the scores of all items. Higher score means better knowledge on dementia.
Change of knowledge on dementia | Knowledge on dementia changes from immediately after intervention to three months after intervention.
  Knowledge on dementia will be assessed by using Dementia Knowledge Assessment Scale. The total score is 0 to 50 by adding up the scores of all items. Higher score means better knowledge on dementia.
Change of attitude towards dementia care | Attitude towards dementia care changes from baseline to immediately after intervention (2 months).
  Attitude towards dementia care will be assessed by using Approaches to Dementia Questionnaire. The total score is 19-95 with higher score indicating the more positive attitudes.
Change of attitude towards dementia care | Attitude towards dementia care changes from immediately after intervention to three months after intervention.
  Attitude towards dementia care will be assessed by using Approaches to Dementia Questionnaire. The total score is 19-95 with higher score indicating the more positive attitudes.
Change of person-centred care approach | Person-centred care approach changes from baseline to immediately after intervention (2 months).
  Person-centred care approach will be assessed by Person-centred care assessment tools. The total score ranges from 15 to 75 with higher score indicating higher degree of person-centred care provision in the institutions.
Change of person-centred care approach | Person-centred care approach changes from immediately after intervention to three months after intervention.
  Person-centred care approach will be assessed by Person-centred care assessment tools. The total score ranges from 15 to 75 with higher score indicating higher degree of person-centred care provision in the institutions.
Change of severity of behavioural and psychological symptoms of dementia (BPSD) of residents with dementia | Severity of BPSD of residents with dementia changes from baseline to immediately after intervention (2 months).
  Severity of BPSD of residents with dementia will be assessed by Neuropsychiatric Inventory - Nursing Home Version (NPI-NH). The frequency × severity of each item yielded a composite symptom, and total severity scores which ranges from 1 to 36 reflecting the sum of each item score. Higher scores indicate more severe symptoms. The total score of caregiver distress range from 12 to 60, with higher score indicating more severe distress.
Change of severity of behavioural and psychological symptoms of dementia (BPSD) of residents with dementia | Severity of BPSD of residents with dementia changes from immediately after intervention to three months after intervention.
  Severity of BPSD of residents with dementia will be assessed by Neuropsychiatric Inventory - Nursing Home Version (NPI-NH). The frequency × severity of each item yielded a composite symptom, and total severity scores which ranges from 1 to 36 reflecting the sum of each item score. Higher scores indicate more severe symptoms. The total score of caregiver distress range from 12 to 60, with higher score indicating more severe distress.
Care staff's satisfaction | Care staff's satisfaction will be measured immediately after the intervention in intervention group.
  Care staff's satisfaction will be measured with a self-developed, five-point Likert, five-item scale including satisfaction with educational content, teaching form, provider, usefulness and overall evaluation. The total score ranges from 5 to 25, with higher score representing more dissatisfaction on the training.

OTHER OUTCOMES:
Participants' experience about the intervention | Focus group interviews will be conducted within one week after the intervention.
  Focus group interviews which will last around 40-60 minutes will be conducted to understand care home staff's experience and their perceptions towards the program.

CONTACTS AND LOCATIONS:
Locations (1):
- 朗诗常青藤养老服务有限公司睿城站, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided